CLINICAL TRIAL: NCT03765112
Title: Macular Involvement in Diabetic Retinopathy Evaluated With Swept-Source OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eduardo Navajas, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H18-02095
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCTA (Experimental): Patients with diabetes and healthy controls will be imaged with optical coherence tomography (OCT) angiography, Spectral domain OCT and ultra wide-field imaging.
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Device: Optical coherence tomography angiography — Multiple scans of the retina will be recorded to evaluate microvascular changes.

SUMMARY:
This study evaluates micro-vascular changes in patients with diabetes. Results of diseased retinas will be compared to healthy controls.

DETAILED DESCRIPTION:
The prevalence of diabetes mellitus (DM) is increasing worldwide. Diabetic retinopathy is the most prevalent complication of DM and a leading cause of visual impairment due to closure of capillaries. High-resolution imaging techniques of the retina and its supplying vascular networks can allow novel insight to subtle changes that cannot be appreciated in standard fundus examination. In this study capillary changes of patients with different severity levels of diabetic retinopathy will be investigated with non-invasive imaging technology to better understand the process of disease progression.

Imaging will be done with Optical Coherence tomography (OCT) angiography as well as spectral domain OCT and ultra wide-field imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 Participants can have 1 or 2 study eyes

Patient Group:

* Diabetes mellitus type 1 or 2
* Study eye with any DR severity level: no DR, mild NPDR, mod NPDR, sev NPDR, PDR

Exclusion Criteria:

* Substantial media opacities that would preclude successful imaging

  * Active intraocular inflammation (grade trace or above) in either eye like infectious conjunctivitis, keratitis, scleritis, endophthalmitis as well as idiopathic or autoimmune-associated uveitis in either eye
  * Structural damage to the center of macula in the study eye
  * History of prior panretinal photocoagulation
  * History of treatment with intravitreal agents over the prior 6 months
  * Macular edema involving the central subfield
  * Prior history of vitrectomy
  * Atrophy of retinal pigment epithelium, subretinal fibrosis, laser scar within foveal avascular zone (FAZ) or organized hard exudate plaques
  * Substantial non-diabetic intraocular pathology in the study eye including retinal vascular occlusion, retinal detachment, macular hole, choroidal neovascularization, macula dystrophies
  * Intraocular surgery (including cataract surgery, YAG laser capsulotomy) in the study eye within 3 months preceding Day 0, or history of corneal transplantation in the study eye
  * Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication)or history of glaucoma filtration surgery
  * Inability to obtain fundus images of sufficient quality to be analyzed and graded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Perfusion density | 6 months
  The density of perfused capillaries (metric variable) measured with optical coherence tomography angiography (OCTA) will be compared between the different severity levels of diabetic retinopathy as well as to the control arm.

SECONDARY OUTCOMES:
Areas of different perfusion density | 6 months
  Perfusion density of the capillary network will be measured at seven different areas and will be compared within the same patient
Foveal avascular zone (FAZ) | 6 months
  Size (area) of FAZ will be compared between the different severity levels of diabetic retinopathy as well as to the control arm.
Foveal avascular zone (FAZ) | 6 months
  The circularity of FAZ will be compared between the different severity levels of diabetic retinopathy as well as to the control arm.
Presence of predominantly peripheral lesions (PPL) | 6 months
  The presence of PPL (categorical variable yes/no) will be correlated with the perfusion density measured with OCTA
Retinal layer thickness | 6 months
  Retinal layer thickness measured with optical coherence tomography (OCT) will be correlated with the perfusion density measured with OCTA
Change in perfusion density in patients with moderate or severe non proliferative diabetic retinopathy (DR) or low risk proliferative DR over the follow up of one year | 18 months
  Patients with moderate or severe non proliferative diabetic retinopathy (DR) or low risk proliferative DR will be followed over one year. Perfusion density will be measured at each timepoint and followed over the year,

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Care Center, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karst SG, Heisler M, Lo J, Schuck N, Safari A, V Sarunic M, Maberley DAL, Navajas EV. Evaluating Signs of Microangiopathy Secondary to Diabetes in Different Areas of the Retina with Swept Source OCTA. Invest Ophthalmol Vis Sci. 2020 May 11;61(5):8. doi: 10.1167/iovs.61.5.8. PMID 32392316